CLINICAL TRIAL: NCT01212692
Title: A Theoretically Based Memory Training Intervention in Mild Cognitive Impairment
Brief Title: Effects of Mental Stimulation in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Paul B. Rosenberg, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00039100; R01AG034934 (NIH)
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mentally stimulating activities (Experimental)
  Interventions: Behavioral: mentally stimulating activities
- Mentally stimulating activities- other (Active Comparator)
  Interventions: Behavioral: mentally stimulating activities

INTERVENTIONS:
Behavioral: mentally stimulating activities — The study will compare the effects of different methods of mental stimulation. The intervention involves 6 classroom-style educational sessions and 10 mental stimulation studies involving computerized memory tasks.

SUMMARY:
The purpose of this study is to learn if activities that challenge the brain (mentally stimulating activities) can improve memory and other types of thinking in patients with Mild Cognitive Impairment. The study will compare the effects of different methods of mental stimulation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years of age
* meet criteria for amnestic-Mild Cognitive Impairment (MCI)
* have capacity to give informed consent
* have capacity to complete assessment measures

Exclusion Criteria:

* history of drug or alcohol dependence
* severe psychiatric conditions associated with psychosis (e.g., schizophrenia)
* recent stroke
* clinical diagnosis of probable Alzheimer's Disease
* history of seizure disorder, serious head trauma, or other medical, psychiatric, or neurological conditions associated with significant cognitive impairment (e.g., Parkinson's Disease, Korsakoff's, HIV)
* current use of Alzheimer's Disease medications (e.g., cholinesterase inhibitors, memantine)

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Self-Ordered Pointing Task | baseline
Trail-Making | baseline
Timed Instrumental Activities of Daily Living | baseline
Rey Auditory Verbal Learning Test | baseline
Self-ordered pointing task | immediately after the intervention
Self-ordered pointing task | 3 months post intervention
Self-ordered pointing task | 9 months post-intervention
Trail-Making | immediately after the intervention
Trail-Making | 3 months post-intervention
Trail-Making | 9 months post-intervention
Timed Instrumental Activities of Daily Living | immediately after the intervention
Timed Instrumental Activities of Daily Living | 3 months post-intervention
Timed Instrumental Activities of Daily Living | 9 months post-intervention
Rey Auditory Verbal Learning Test | immediately after the intevention
Rey Auditory Verbal Learning Test | 3 months post-intervention
Rey Auditory Verbal Learning Test | 9 months post-intervention

SECONDARY OUTCOMES:
Clinical Dementia Rating Scale | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Digit Symbol Substitution Test | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Digit Span | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Verbal Fluency Test | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Geriatric Depression Scale | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Neuropsychiatric Inventory | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Recollection Task | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
N-Back | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Rivermead Behavioral Memory Test | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Instrumental Activities of Daily Living | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Functional Capacities for Activities of Daily Living | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention
Multifactorial Memory Questionnaire | baseline, immediately after the intervention, 3 months post intervention, and 9 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Rosenberg, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- BPRU, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States